CLINICAL TRIAL: NCT04501731
Title: Controlling Coordination After Childhood Cerebellar Cancer - Pilot Study
Brief Title: Controlling Coordination After Childhood Cerebellar Cancer, a Pilot Study
Acronym: 5C-pilot
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospital NHS Trust (Unknown); Nottingham Hospitals Charity (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20047
Record Dates: First submitted 2020-07-23; First posted 2020-08-06 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2021-09

CONDITIONS: Brain Cancer
Keywords: Motor recovery; Transcranial Magnetic Stimulation; Magnetic Resonance Imaging; Paediatric; Cerebellum; Posterior Fossa Tumour
MeSH Terms: conditions — Brain Neoplasms | interventions — Transcranial Magnetic Stimulation; Magnetic Resonance Spectroscopy; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young PFT survivors
  Interventions: Other: Transcranial Magnetic Stimulation (TMS); Other: Magnetic Resonance Imaging (MRI); Other: Motor assessment; Other: Questionnaires
- Age-matching controls
  Interventions: Other: Transcranial Magnetic Stimulation (TMS); Other: Magnetic Resonance Imaging (MRI); Other: Motor assessment

INTERVENTIONS:
Other: Transcranial Magnetic Stimulation (TMS) — With the TMS session we gather information about nerve fibres from the brain to the hand. It will last around 2 hours and 30 minutes.
Other: Magnetic Resonance Imaging (MRI) — With the MRI scan we will gather information about the brain structure and function. This will last around 30 minutes.
Other: Motor assessment — The motor assessment includes a pegboard game, a "grab the alien nose" game and measure of your maximum grip force. In total it will last around 30 minutes.
Other: Questionnaires — Feasibility, tolerability of such intervention as well as quality of life of PFT survivors will be assessed thanks to questionnaires.
  Groups: Young PFT survivors

SUMMARY:
Posterior fossa tumours (PFT) account for 2/3 of childhood brain cancers. They can be highly malignant requiring combined chemotherapy and radiotherapy post-surgery for a >50% chance of cure. PFT frequently involve the cerebellum which is responsible for coordinating movement, balance, emotional control, and links closely to control of affect and executive function. PFT survivors show highly variable profiles for cognitive and sensorimotor functioning which are influenced strongly by the severity of the pre-diagnostic or post-surgical brain injury

State-of-the-art magnetic resonance imaging (MRI) scans can allow to measure a variety of different biological processes in the brain, and the investigators believe that some of these MRI measures (called MRI biomarkers) have the potential to improve our ability to understand and monitor consequences of the ablative brain surgery and complex mechanisms of motor skills recovery. Biomarkers are very important for the development of intervention because 1) they help understand the recuperation process and 2) they allow to effectively assess whether or not a treatment or intervention works.

Transcranial magnetic stimulation (TMS) is a powerful non-invasive neuro-modulatory intervention that has the potential to evaluate the integrity of the nervous tracts from the brain to the hand. It is a procedure that applies magnetic pulses on the surface of the scalp to reach underlying brain tissue. TMS has built a reputable status among neuro-rehabilitative research, and there is currently a major effort to translate the positive research findings into clinically useful therapeutic strategies.

This study is therefore an important first step towards understanding how potential MRI biomarkers and responses to TMS relate to motor symptoms in PFT young survivors. Once completed, this study will allow the investigators to select the most promising MRI biomarkers and TMS protocols to take forward into future treatment trials. The investigators aim to stimulate the recovery of coordination skills, help the development of targeted therapies, and consequently improve long-term quality of life in children and young people with history of brain tumour.

The proposed research intends to prove the feasibility of such brain stimulation and imaging and collect some preliminary measures

ELIGIBILITY:
Inclusion Criteria:

* Able to undergo MRI scan without sedation or general anaesthetic
* Able to give informed consent.

Exclusion Criteria:

* History of seizure
* Current cancer or post surgery treatment
* Contraindication to TMS or MRI
* Pregnancy

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 4 participants with history of PFT (no history of seizure, no current cancer treatment) 6 healthy controls (no history of brain injury)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
5C-pilot Satisfaction Questionnaire | 6 months
  Participants rating their experience of MRI, TMS and motor assessment
Completion rate of the sessions of TMS, MRI and motor tasks | 6 months
  Measure of quality of MRI images (participants motion) - Feasibility will be confirmed if 50% or more of these participants complete the TMS session

SECONDARY OUTCOMES:
Anatomical MRI metrics (PFT vs control) | 1 year
  Cerebellar volumetry and cerebellar parcellation - after surgery (mm3)
fMRI metrics (PFT vs control) | 1 year
  Functional connectivity within sensorimotor network (activation map)
Diffusion MRI metrics (PFT vs control) | 1 year
  Anatomical connectivity within sensorimotor network (tractography)
Single-pulse TMS metrics (PFT vs control) | 1 year
  Resting motor threshold (Stimulus intensity expressed as a percentage of maximal stimulator output)
Single-pulse TMS metrics (PFT vs control) | 1 year
  input-output curve
Single-pulse TMS metrics (PFT vs control) | 1 year
  Silent period (ms)
Single-pulse TMS metrics (PFT vs control) | 1 year
  Short-afferent inhibition
Dual-pulse TMS metrics (PFT vs control) | 1 year
  Intracortical & long-latency inhibition and facilitation
Dual-pulse TMS metrics (PFT vs control) | 1 year
  cerebellar-motor inhibition
Motor performance (PFT vs control) - Reaching and grasping task | 1 year
  Kinematic parameters of movement
Motor performance (PFT vs control) - Grooved pegboard | 1 year
  Score
Motor performance (PFT vs control) - Grip force | 1 year
  Maximum force (N)
Quality of life of PFT survivors: FACT-Peds-Br Questionnaire | 6 months
  FACT-Peds-Br Pediatric Questionnaire - For patients with Brain cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's Medical Centre, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided